CLINICAL TRIAL: NCT02751424
Title: A Phase I, Randomized, Double-Blind (Sponsor Unblinded), Single-Center, Placebo-Controlled, Two-Part Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Ascending Single and Repeat Intravenous Doses of GSK3342830 in Healthy Adult Subjects
Brief Title: A Study to Evaluate Safety, Tolerability and Pharmacokinetics of Ascending Intravenous Single Dose and Repeat Dose of GSK3342830
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study data is currently under review.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 204847
Record Dates: First submitted 2016-04-21; First posted 2016-04-26 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-06

CONDITIONS: Infections, Bacterial
Keywords: Multidrug-resistant; Gram negative bacterial infection; Safety; Pharmacokinetic
MeSH Terms: conditions — Bacterial Infections; Gram-Negative Bacterial Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK3342830 single dose in Part 1 (Experimental): Enrolled subject will receive single escalation dose of GSK3342830. The escalating doses will be evaluated in six cohorts as A- 250 mg, B-500 mg, C-1000 mg, D-2000 mg, E-4000 mg, and F-=<6000 mg. In each cohort 6 subjects will receive GSK3342830 in form of infusion for 1 h, therefore approximately 36 subjects will receive GSK3342830. Dose escalation will be based on evaluation of the preceding dose levels in the study.
  Interventions: Drug: GSK3342830
- Placebo single dose in Part 1 (Placebo Comparator): Enrolled subject will receive single escalation dose of placebo. In each cohort, 2 subjects will receive placebo in form of infusion for 1 h, therefore approximately 12 subjects will receive placebo.
  Interventions: Drug: Placebo
- GSK3342830 repeat Dose in Part 2 (Experimental): Enrolled subject will receive repeat escalating dose of GSK3342830. GSK3342830 as a single IV infusion will be administered on Day 1, TID (8 hours apart) IV infusions on Days 2 through 14, and a single IV infusion on Day 15. The escalating doses will be evaluated in three cohorts as G-1000 mg, H-2000 and I-4000 mg. In each cohort 8 subjects will receive GSK3342830 in form of infusion for 1 h, therefore approximately 24 subjects will receive GSK3342830. The starting dose and maximum dose may change based on clinical safety and PK findings in Part 1 or earlier doses in Part 2 respectively.
  Interventions: Drug: GSK3342830
- Placebo repeat Dose in Part 2 (Placebo Comparator): Enrolled subject will receive repeat escalation dose of placebo. Placebo as a single IV infusion will be administered on Day 1, TID (8 hours apart) IV infusions on Days 2 through 14, and a single IV infusion on Day 15. In each cohort, 2 subjects will receive placebo in form of infusion for 1 h, therefore approximately 6 subjects will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3342830 — A pyrogen free lyophilized formulation, white to yellowish brown powder containing 1000 mg of GSK3342830A (as free base) per vial. The reconstituted solution looks like a clear, colorless to yellow or brownish yellow liquid, free from visible particulate matter will be administered as IV infusion over 1 hour.
  Arms: GSK3342830 repeat Dose in Part 2; GSK3342830 single dose in Part 1
Drug: Placebo — A clear and colorless solution containing 0.9% sodium chloride. It will administered as IV infusion over 1 hour.
  Arms: Placebo repeat Dose in Part 2; Placebo single dose in Part 1

SUMMARY:
A phase I, first-time-in-human (FTIH), randomized, double-blind, placebo controlled, dose-escalation study is conducted to determine the safety, tolerability, and pharmacokinetic (PK) profile of GSK3342830 after administration of single intravenous (IV) infusion in Part 1 and repeat IV infusion in Part 2 in healthy subjects. Part 1 will investigate escalating single IV doses of GSK3342830. Part 2, will investigate escalating repeat IV doses of GSK3342830 with repeat dosing for 15 days as follows: a single IV infusion on Day 1, TID (three times a day) IV infusions on Days 2 through 14 (approximately every 8 hours), and a single IV infusion on Day 15. The planned starting GSK3342830 dose in Part 1 is 250 milligram (mg) administered as a single IV infusion. The dose is planned to increase in subsequent cohorts to 500, 1000, 2000, 4000, and less than or equal to (≤) 6000 mg. Part 1 will be divided into 6 cohorts (A-F) and each cohort will enroll 10 subjects (6 in active and 2 in placebo). Dose escalation will be conducted only if it is supported by the preliminary safety, tolerability, and PK results from the preceding dose levels in the study. The repeat dose escalation component (Part 2) of this study will be planned to be initiated after completion and evaluation of the all single dose cohorts up to and including 4000 mg.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age, inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter outside the reference range for the population being studied may be included only if the investigator feels and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >50 kilogram (kg) (110 pounds [lb]) for men and >40 kg (99 lb) for women and body mass index within the range of 18.5 to 30 kg per square meter (m^2), inclusive.
* Male or Female subjects. Males: Male subjects with female partners of child-bearing potential must agree to use one of the highly effective contraception from the time of first dose of study drug until completion of the Follow-up visit, and Females: A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotropin [hCG] test), not lactating, and considered to be of non-reproductive potential (non-reproductive potential is defined as: Pre-menopausal females with one of the following: Documented tubal ligation or Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion or Hysterectomy or Documented bilateral oophorectomy).
* Postmenopausal defined as 12 months of spontaneous amenorrhea and in questionable cases a blood sample with simultaneous follicle-stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels)
* Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods, if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post menopausal status before study enrolment.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions.

Exclusion Criteria:

* Alanine aminotransferase (ALT) not within normal limits; bilirubin >1.5× upper limit of normal (ULN; isolated bilirubin >1.5× ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Corrected QT (QTc) >450 milliseconds (msec).
* Any clinically significant central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic, or gastrointestinal condition or history of such a condition that, in the opinion of the investigator, may place the subject at an unacceptable risk as a participant in this trial or may interfere with the absorption, distribution, metabolism, or excretion of drugs.
* Use of a systemic antibiotic within 30 days of screening.
* Ongoing febrile illness.
* Confirmed history of Clostridium difficile diarrhea
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before the first dose of study treatment, unless in the opinion of the Investigator, the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of screening defined as an average weekly intake of >21 units (or an average daily intake of >3 units) for males or an average weekly intake of >14 units (or an average daily intake >2 units) for females. One unit is equivalent to 270 milliliter (mL) of full strength beer, 470 mL of light beer, 30 mL of spirits, or 100 mL of wine.
* Urinary cotinine level indicative of smoking or history or regular use of tobacco- or nicotine containing products within 3 months before screening.
* History of hypersensitivity attributed to beta-lactam antibiotics (including cephalosporin, carbapenem, or penicillin antibiotics) or other drugs, a history of multiple antibiotic intolerances, or a history of serious adverse drug reactions.
* Sensitivity to poison ivy or other catechol-related hypersensitivity (e.g., mango allergy).
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of latex allergy.
* History of sensitivity to any of the study treatments or components thereof, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation in the study.
* Presence of hepatitis B surface antigen or positive hepatitis C antibody test result at screening or within 3 months before the first dosing day in this study.
* Serum creatinine >ULN.
* Glomerular filtration rate <90 millilter per minute per 1.73 square meter (mL/min/1.73m^2) as calculated by the Chronic Kidney Disease Epidemiology Collaboration formula
* Albumin to creatinine ratio (ACR) >0.03 mg/mg. In the event of an ACR above this threshold, eligibility may be confirmed by a second measurement.
* Urinalysis positive for blood without other cause identified.
* A positive pre-study drug or alcohol screen.
* A positive test for human immunodeficiency virus antibody at or before screening.
* Participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period before the first dosing day in this study: 30 days, 5 half lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 new chemical entities within 12 months before the first dosing day in this study.
* Exclusion criteria for screening and baseline 12-lead ECG: Heart rate <40 and >100 beats per minute for males and <50 and >100 beats per minute (for females), pulse rate is <120 and >220 msec, QRS is <70 and >120 msec, and corrected QT interval using Bazett's formula (QTcB ) and corrected QT interval using Fridericia's formula (QTcF ) >450 msec.. Also apart from this, subject having evidence of previous myocardial infarction, bundle branch block and Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolf-Parkinson-White syndrome), sinus pauses more than 3 seconds, non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats), or any significant arrhythmia that, in the opinion of the investigator will interfere with the safety of the individual subject.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Adelaide, South Australia, Australia

REFERENCES:
- [Derived] Tenero D, Farinola N, Berkowitz EM, Tiffany CA, Qian Y, Xue Z, Raychaudhuri A, Gardiner DF. Pharmacokinetics, Safety, and Tolerability Evaluation of Single and Multiple Doses of GSK3342830 in Healthy Volunteers. Clin Pharmacol Drug Dev. 2019 Aug;8(6):754-764. doi: 10.1002/cpdd.637. Epub 2018 Dec 10. PMID 30536589

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a first-time-in-human (FTIH), randomized, double-blind, placebo-controlled, dose-escalation study to determine the safety, tolerability & pharmacokinetic (PK) profile of GSK3342830 after administration of single (Part 1) & repeat (Part 2) IV doses in healthy adult participants (par.) & single IV dose in healthy adult Japanese par. (Part 3).
Pre-assignment Details: A total of 62 par. were enrolled in the study. Part 1 comprised of 48 par. and 14 par. were enrolled in Part 2. No par. were enrolled in Part 3 as the study was terminated early per sponsor discretion.
Groups:
- GSK3342830 250 mg: Healthy adult participants in this cohort, were administered GSK3342830 dose in Part 1 as 250 milligram (mg),for 1 hour (hr) as a single intravenous (IV) infusion, on Day 1.
- GSK3342830 500 mg: Healthy adult participants in this cohort received an escalated dose GSK3342830 at 500 mg, for 1 hr, as a single IV infusion on Day 1.
- GSK3342830 1000 mg: The healthy adult participants in this cohort received an escalated dose GSK3342830 at 1000 mg, for 1 hr, as a single IV infusion on Day 1.
- GSK3342830 2000 mg: The healthy adult participants in this cohort received an escalated dose of GSK3342830 at 2000 mg, for 1 hr, as a single IV infusion on Day 1.
- GSK3342830 4000 mg: The healthy adult participants in this cohort received an escalated dose of GSK3342830 at 4000 mg, for 1 hr, as a single IV infusion on Day 1.
- GSK3342830 6000 mg: The healthy adult participants in this cohort received an escalated dose of GSK3342830 at 6000 mg, for 1 hr, as a single IV infusion on Day 1.
- Placebo, Part 1: Healthy adult participants from each cohort received placebo in form of infusion for 1 hr, on Day 1.
- GSK3342830 1000 mg TID: Healthy adult participants in this repeat dose escalation cohort were administered GSK3342830 dose, in Part 2 as 1000 mg, as a single IV infusion on Day 1, three times a day (TID) IV infusions (approximately every 8 hrs) on Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14, and a single IV infusion on Day 15.
- Placebo, Part 2: Healthy adult participants in this repeat dose escalation cohort were administered with matching placebo to GSK3342830 1000 mg TID, Single IV infusion on Day 1, TID IV infusions (approximately every 8 hrs) on Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14, and a single IV infusion on Day 15.
Period: Part 1
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg | Placebo, Part 1 | GSK3342830 1000 mg TID | Placebo, Part 2
Started | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 0 | 0
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg | Placebo, Part 1 | GSK3342830 1000 mg TID | Placebo, Part 2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK3342830 250 mg: Healthy adult participants in this cohort, were administered GSK3342830 dose in Part 1 as 250 mg, for 1 hr as a single IV infusion, on Day 1.
- GSK3342830 1000 mg TID: Healthy adult participants in this repeat dose escalation cohort were administered GSK3342830 dose, in Part 2 as 1000 mg, as a single IV infusion on Day 1, TID IV infusions (approximately every 8 hrs) on Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14, and a single IV infusion on Day 15.
- Total: Total of all reporting groups
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg | Placebo, Part 1 | GSK3342830 1000 mg TID | Placebo, Part 2 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 11 | 3 | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.2 (3.54) | 22.8 (2.64) | 32.2 (10.57) | 25.5 (3.78) | 30.2 (7.70) | 21.0 (1.10) | 28.3 (5.68) | 27.1 (3.99) | 22.3 (1.53) | 26.4 (6.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 11 | 3 | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 5 | 4 | 5 | 4 | 6 | 10 | 10 | 2 | 52
  Black or African American | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 4
  Asian | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 6
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Multiple | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Adverse Event (AE) and Serious Adverse Event (SAE)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, Requires hospitalization or prolongation of existing hospitalization, Results in disability/incapacity, Is a congenital anomaly/birth defect, medical judgement and is associated with liver injury or liver impartment. The number of participants with AEs and SAEs assessed in Part 1 (Single dose) of the study were reported.
Time Frame: Up to Day 43
Population: Safety population comprised of all participants who received at least 1 dose of study drug and had at least one post-dose safety assessment.
Measure: Number; unit: Participants
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg | Placebo, Part 1
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
Participants
  Any AE | 5 | 4 | 6 | 5 | 5 | 4 | 11
  Any SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part 2: Number of Participants With AE and SAE
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, Requires hospitalization or prolongation of existing hospitalization, Results in disability/incapacity, Is a congenital anomaly/birth defect, medical judgement and is associated with liver injury or liver impartment. The number of participants with AEs and SAEs assessed in Part 2 (Repeat dose) of the study were reported.
Time Frame: Up to Day 56
Population: Safety population.
Measure: Number; unit: Participants
Groups:
- GSK3342830 1000 mg TID: Healthy adult participants in this repeat dose escalation cohort were administered GSK3342830 dose, in Part 2 as 1000 mg, as a single IV infusion on Day 1, TID, IV infusions (approximately every 8 hrs) on Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14, and a single IV infusion on Day 15.
Arm/Group | GSK3342830 1000 mg TID | Placebo, Part 2
Number analyzed (Participants) | 11 | 3
Participants
  Any AE | 11 | 3
  Any SAE | 0 | 0

3. Primary Outcome: Part 1: Number of Participants With Abnormal Hematology Parameters as a Measure of Safety-Grade 3 or Higher
Description: Blood samples were collected and processed to measure the number of participants with abnormal platelet counts, red blood cells (RBC) count, white blood cells (WBC) count (absolute), hemoglobin, hematocrit, reticulocytes, total iron, total iron binding capacity (TIBC), ferritin, RBC indices (mean corpuscle volume [MCV], mean corpuscle hemoglobin [MCH] and mean corpuscle hemoglobin concentration [MCHC]) and differential WBC count (neutrophils, lymphocytes, monocytes, eosinophil's, and basophils). Participants with abnormalities of Grade 3 or higher have been reported.
Time Frame: Up to Day 2
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg | Placebo, Part 1
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part 2: Number of Participants With Abnormal Hematology Parameters as a Measure of Safety-Grade 3 or Higher
Description: Blood samples were collected and processed to measure the number of participants with abnormal platelet counts, RBC count, WBC count (absolute), hemoglobin, hematocrit, reticulocytes, total iron, TIBC, ferritin, RBC indices MCV, MCH and MCHC and differential WBC count (neutrophils, lymphocytes, monocytes, eosinophils, and basophils). These were collected on Day 2, 5, 10 and Day 15, during Part 2 of the study. Part 2 is repeat dose escalation. Participants with abnormalities of Grade 3 or higher have been reported.
Time Frame: Up to Day 15
Population: Safety population.
Measure: Number; unit: Participants
Arm/Group | GSK3342830 1000 mg TID | Placebo, Part 2
Number analyzed (Participants) | 11 | 3
Participants | 0 | 0

5. Primary Outcome: Part 1: Number of Participants With Abnormal Clinical Chemistry Parameters as a Measure of Safety-Grade 3 or Higher
Description: Blood samples were collected and processed to measure the number of participants with abnormal blood urea nitrogen (BUN), creatinine, glucose, bicarbonate, sodium, potassium, chloride, calcium, aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT), alkaline phosphatase (ALP) levels, uric acid, total and direct bilirubin, total protein and albumin. These were collected on Day 1, during Part 1(single dose escalation) of the study. Participants with abnormalities Grade 3 or higher were reported.
Time Frame: Day 2
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg | Placebo, Part 1
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part 2: Number of Participants With Abnormal Clinical Chemistry Parameters as a Measure of Safety-Grade 3 or Higher
Description: Blood samples were collected and processed to measure the number of participants with abnormal BUN, creat, glucose, bicarbonate, sodium, potassium, chloride, calcium, AST/SGOT, ALT/SGPT, ALP levels, uric acid, total and direct bilirubin, total protein and albumin. These were collected on Day 2, 5, 10 and Day 15 during Part 2 (repeat dose escalation), of the study. Participants with abnormalities Grade 3 or higher were reported.
Time Frame: Up to Day 15
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | GSK3342830 1000 mg TID | Placebo, Part 2
Number analyzed (Participants) | 11 | 3
Participants
  Serum Glucose | 1 | 0
  Serum or Plasma ALT | 1 | 0
  Serum or Plasma albumin | 1 | 0
  Serum or Plasma ALP | 0 | 0
  Serum or Plasma AST | 2 | 0
  Serum or Plasma Calcium | 0 | 0
  Serum or Plasma Chloride | 0 | 0
  Serum or Plasma Creat | 0 | 0
  Serum or Plasma Direct Bilirubin | 2 | 0
  Serum or Plasma Potassium | 1 | 0
  Serum or Plasma Protein | 0 | 0
  Serum or Plasma Sodium | 1 | 0

7. Primary Outcome: Part 1: Number of Participants Having Abnormal Urine Parameters (Using Dipstick Test) as a Measure of Safety
Description: An aliquot of the urine samples from first morning void urine samples was collected to analyze specific gravity, pH, glucose, protein, blood and ketone bodies by dipstick method, microscopic examination (if blood or protein is abnormal), albumin to creatinine ration (ACR), neutrophil gelatinase associated lipocalin (NGAL) and kidney injury molecule-1 (KIM-1). Urine samples were analyzed after the end of the study to verify if a clinical signal is detected. Urine samples were collected on Day 1 of Part 1 (Single-dose escalation) of the study.
Time Frame: Up to Day 2
Population: Safety population.
Measure: Number; unit: Participants
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg | Placebo, Part 1
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Part 2: Number of Participants Having Abnormal Urine Parameters (Using Dipstick Test) as a Measure of Safety
Description: An aliquot of the urine samples from first morning void urine samples was collected to analyze specific gravity, pH, glucose, protein, blood and ketone bodies by dipstick method, microscopic examination (if blood or protein is abnormal), ACR, NGAL and KIM-1. These urine samples were analyzed after the end of the study to verify if a clinical signal is detected. The samples were collected on Day 2, 5, 10, and Day 15 of Part 2 (Repeat dose escalation) of the study.
Time Frame: Day 2, 5, 10 and Day 15
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | GSK3342830 1000 mg TID | Placebo, Part 2
Number analyzed (Participants) | 11 | 3
Participants | 0 | 0

9. Primary Outcome: Part 1: Number of Participants With Electrocardiogram (ECG) Parameters of Potential Clinical Importance (PCI)
Description: Triplicate 12-lead ECGs were obtained at least 5 minutes apart within 1 hr before dosing. Single ECGs were obtained at all other time points on Day 1 at 0.5 hr, 1 hr, 1.5 hr, 2, 3, 4, 6, 12 and 24 hr, Day 2 (36 hr) and Day 3 (48 hr) during Part 1 (single dose escalation phase) of the study. All the 12-lead ECGs were measured using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals.
Time Frame: Up to Day 3
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg | Placebo, Part 1
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
Participants
  Heart Rate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR Interval | 0 | 1 | 0 | 0 | 0 | 0 | 0
  QRS Duration | 0 | 0 | 1 | 3 | 1 | 1 | 2
  QT Interval | 1 | 2 | 1 | 0 | 0 | 1 | 2
  QTc (Bazett) | 1 | 1 | 1 | 1 | 2 | 2 | 3
  QTc (Fridericia) | 1 | 0 | 1 | 0 | 1 | 0 | 1
  RR Interval | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Part 2: Number of Participants With ECG Parameters of PCI
Description: Triplicate 12-lead ECGs were obtained at least 5 minutes apart within 1 hr before the start of infusion (pre-dose) on Day 1. Single ECGs were obtained at 0.5, 1, 1.5, 2, 3, 4, 6, and 12 hrs after the start of infusion on Day 1 and Day 15, within 1 hr before the start of the morning infusion on Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14, and in the morning on Day 16. All the 12-lead ECGs were measured using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals.
Time Frame: Up to Day 16
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | GSK3342830 1000 mg TID | Placebo, Part 2
Number analyzed (Participants) | 11 | 3
Participants
  Heart Rate | 0 | 0
  PR Interval | 1 | 0
  QRS Duration | 0 | 0
  QT Interval | 1 | 2
  QTc (Bazett) | 2 | 1
  QTc (Fridericia) | 1 | 1
  RR Interval | 0 | 0

11. Primary Outcome: Part 1: Number of Participants With Vital Signs of Potential Clinical Importance (PCI)
Description: The vital sign includes systolic blood pressure, diastolic blood pressure, heart rate, respiratory rate and temperature which were measured in a semi-supine position, where the participant had rested in the same position for at least 5 minutes. The number of participants with vital values, of PCI were reported. These were collected on Day 1 at pre-dose, 0.5 hr, 1 hr, 1.5 hr, 2, 3, 4, 6, 12 and 24 hr, Day 2 (36 hr) and Day 3 (48 hr) during Part 1 (single dose escalation phase) of the study.
Time Frame: Up to Day 3
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg | Placebo, Part 1
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
Participants
  Systolic Blood Pressure | 1 | 0 | 0 | 1 | 0 | 0 | 1
  Diastolic Blood Pressue | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Pulse rate | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Temperature | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory rate | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Part 2: Number of Participants With Vital Signs of PCI
Description: The vitals for systolic, diastolic blood pressure, heart rate, respiratory rate and temperature were taken in a semi-supine position, where the participant had rested in the same position for atleast 5 minutes. The number of participants with vital values, of PCI were reported. These were collected from Day 1 to Day 16. Assessments were done within 1 hr before the start of infusion (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, and 12 hrs after the start of infusion on Days 1 and 15, within 1 hr before the start of the morning infusion and on Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14, and in the morning on Day 16.
Time Frame: Up to Day 16
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | GSK3342830 1000 mg TID | Placebo, Part 2
Number analyzed (Participants) | 11 | 3
Participants
  SBP | 0 | 0
  DBP | 0 | 1
  Pulse rate | 1 | 0
  Temperature | 0 | 0
  Respiratory rate | 0 | 0

13. Secondary Outcome: Part 1-Area Under the Plasma Concentration (AUC) From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration Across All Treatments AUC(0-t) for GSK3342830
Description: AUC (0-t) is defined as AUC from time zero to the last quantifiable concentration after dosing. Blood samples were collected on Day 1 at indicated timepoints (pre-dose, 0.5 hr, 1hr, 1.25 hr, 1.5 hr, 2 hr, 3 hr,3.5 hr, 4 hr, 4.5 hr, 5 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr 24 hr, 36 hr and 48 hr post-dose. The Part 1 phase of the study comprised of single dosing of participants. Log untransformed values for AUC (0-t) have been presented.
Time Frame: Day 1 (pre-dose, 0.5 hr, 1 hr, 1.25 hr, 1.5 hr, 2 hr, 3 hr, 3.5 hr, 4 hr, 4.5 hr, 5 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr, 24 hr, 36 hr, 48 hr post-dose
Population: The Pharmacokinetic (PK) Parameter Population included all participants in the PK population for whom valid and evaluable PK parameters were derived. PK Population is defined as all participants who received at least 1 dose of GSK3342830 and have evaluable PK data for GSK3342830.
Measure: Mean (Standard Deviation); unit: hour *microgram per milliliter
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hour *microgram per milliliter | 40.24 (5.9451) | 93.92 (11.849) | 171.3 (28.299) | 344.0 (30.312) | 672.9 (99.383) | 1039 (134.97)

14. Secondary Outcome: Part 1-AUC Pre Dose to Infinite (Inf) Time (AUC [0-inf]) of GSK3342830
Description: AUC (0-inf) is defined as AUC extrapolated from time zero to infinity. Blood samples were collected on Day 1 at indicated timepoints pre-dose, 0.5 hr, 1hr, 1.25 hr, 1.5 hr, 2 hr, 3 hr,3.5 hr, 4 hr, 4.5 hr, 5 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr 24 hr, 36 hr and 48 hr post-dose. This part 1 phase of the study comprised of single dosing of the participants. Log untransformed values for AUC (0-inf) have been presented.
Time Frame: Day 1 (pre-dose, 0.5 hr, 1 hr, 1.25 hr, 1.5 hr, 2 hr, 3 hr, 3.5 hr, 4 hr, 4.5 hr, 5 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr, 24 hr, 36 hr, 48hr post-dose
Population: PK Parameter Population
Measure: Mean (Standard Deviation); unit: hour *microgram per milliliter
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hour *microgram per milliliter | 42.08 (14.6) | 95.76 (12.5) | 172.5 (15.9) | 346.0 (9.2) | 671.6 (14.5) | 1038 (12.6)

15. Secondary Outcome: Part 1-Maximum Plasma Concentration (Cmax) of GSK3342830
Description: Cmax was defined as the maximum concentration of drug GSK3342830, in plasma. Blood samples were collected on Day 1 at indicated timepoints pre-dose, 0.5 hr, 1hr, 1.25 hr, 1.5 hr, 2 hr, 3 hr,3.5 hr, 4 hr, 4.5 hr, 5 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr 24 hr, 36 hr and 48 hr post-dose. This part 1 phase of the study comprised of single dosing of the participants. Log untransformed values for Cmax have been presented.
Time Frame: as for outcome 13
Population: PK Parameter Population
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Microgram per milliliter | 16.37 (2.9161) | 35.09 (5.8409) | 71.11 (11.109) | 117.4 (41.338) | 242.4 (31.907) | 389.8 (31.010)

16. Secondary Outcome: Part 1-Time to Maximum Plasma Concentration (Tmax) of GSK3342830
Description: Tmax was defined as time required to achieve Cmax for drug GSK3342830, in plasma. Blood samples were collected on Day 1 at indicated timepoints pre-dose, 0.5 hr, 1hr, 1.25 hr, 1.5 hr, 2 hr, 3 hr,3.5 hr, 4 hr, 4.5 hr, 5 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr 24 hr, 36 hr and 48 hr post-dose. This part 1 phase of the study comprised of single dosing of the participants. Log untransformed values for tmax have been presented.
Time Frame: as for outcome 14
Population: PK Parameter Population.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hour | 1.042 (0.1021) | 1.000 (0.0000) | 1.000 (0.0000) | 1.167 (0.4082) | 1.000 (0.0000) | 1.000 (0.0000)

17. Secondary Outcome: Part 1-Terminal Elimination Half-life (t1/2) of GSK3342830 in Plasma
Description: t ½ is defined as the time required by the drug to reduce to half its quantity. Blood samples were collected on Day 1 at indicated timepoints pre-dose, 0.5 hr, 1hr, 1.25 hr, 1.5 hr, 2 hr, 3 hr,3.5 hr, 4 hr, 4.5 hr, 5 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr 24 hr, 36 hr and 48 hr post-dose. This part 1 phase of the study comprised of single dosing of the participants. Log untransformed values for t1/2 have been presented.
Time Frame: as for outcome 13
Population: PK Parameter Population
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hour | 1.860 (0.19150) | 2.139 (0.30026) | 2.295 (0.22578) | 2.596 (0.34939) | 2.465 (0.33519) | 2.461 (0.33327)

18. Secondary Outcome: Part 1-Total Systemic Clearance (CL) of GSK3342830 in Plasma
Description: The systemic CL is a PK measure of volume of plasma from which the drug is removed per unit time. Blood samples were collected on Day 1 at indicated timepoints pre-dose, 0.5 hr, 1hr, 1.25 hr, 1.5 hr, 2 hr, 3 hr,3.5 hr, 4 hr, 4.5 hr, 5 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr 24 hr, 36 hr and 48 hr post-dose. This part 1 phase of the study comprised of single dosing of the participants. Log untransformed values for CL have been presented.
Time Frame: as for outcome 13
Population: PK Parameter Population
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Liter per hour | 5.994 (0.88869) | 5.255 (0.63134) | 5.857 (0.90413) | 5.801 (0.55138) | 6.007 (0.85700) | 5.819 (0.70924)

19. Secondary Outcome: Part 1-Steady-state Volume (Vss) of Distribution of GSK3342830 in Plasma
Description: Vss reflects the actual blood and tissue volume into which a drug is distributed and the relative binding of drug to protein in these spaces. Blood samples were collected on Day 1 at indicated timepoints pre-dose, 0.5 hr, 1hr, 1.25 hr, 1.5 hr, 2 hr, 3 hr,3.5 hr, 4 hr, 4.5 hr, 5 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr 24 hr, 36 hr and 48 hr post-dose. This part 1 phase of the study comprised of single dosing of the participants. Log untransformed values for Vss have been presented.
Time Frame: as for outcome 13
Population: PK Parameter Population
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Liter | 14.65 (2.6449) | 13.98 (2.2987) | 15.54 (2.4329) | 19.87 (11.115) | 16.63 (1.2716) | 15.61 (1.3961)

20. Secondary Outcome: Part 1-Urinary Excretion Ratio Relative to Dose (Feu [t1-t2]) of GSK3342830
Description: Urine samples were collected at indicated timepoints pre-dose and post dose. The Feu has been reported from 0 to 4, 4 to 8, 8 to 12, 12 to 24 and 24 to 48 hrs. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data is not available. The standard deviation could not be calculated as only single participant was present. Log untransformed values for Feu (t1-t2) have been presented.
Time Frame: as for outcome 13
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Percentage of excretion ratio
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Percentage of excretion ratio
  Feu (0-4) (n=6,6,6,6,6,6) | 68.66 (10.456) | 83.01 (49.110) | 71.85 (23.591) | 59.29 (21.740) | 68.39 (5.8313) | 73.42 (8.3037)
  Feu (4-8) (n=6,6,6,6,6,6) | 21.38 (6.2577) | 21.52 (2.7078) | 18.00 (4.3264) | 20.44 (1.3961) | 22.33 (7.1655) | 19.11 (2.5950)
  Feu (8-12) (n=6,6,6,6,6,6) | 3.612 (0.48583) | 4.627 (1.0872) | 4.794 (0.68561) | 6.861 (3.7957) | 5.102 (1.5791) | 5.336 (1.9488)
  Feu (12-24) (n=6,6,6,6,6,6) | 2.173 (1.0482) | 2.557 (0.68228) | 2.039 (0.82840) | 3.967 (4.3285) | 1.972 (1.0979) | 1.941 (0.91904)
  Feu (24-48) (n=1,1,6,6,6,6): number analyzed (Participants) | 1 | 1 | 6 | 6 | 6 | 6
  Feu (24-48) (n=1,1,6,6,6,6) | 0.2132 (NA) — NA indicates that data is not available. The standard deviation could not be calculated as only single participant was present. | 0.2371 (NA) — NA indicates that data is not available. The standard deviation could not be calculated as only single participant was present. | 0.2036 (0.038871) | 0.2245 (0.067861) | 0.1720 (0.069232) | 0.1809 (0.057906)

21. Secondary Outcome: Part 1-Renal Clearance (CLr) of GSK3342830 in Urine
Description: The renal clearance (CLr) is a PK measure of volume of drug is removed per unit time. Urine samples were collected at indicated timepoints pre-dose and post dose. This part 1 phase of the study comprised of single dosing of the participants. Log untransformed values for CLr have been presented.
Time Frame: as for outcome 14
Population: PK Parameter Population
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Liter per hour | 5.709 (0.97041) | 5.696 (1.9452) | 5.771 (2.0146) | 5.229 (0.32521) | 5.867 (0.70267) | 5.837 (0.98448)

22. Secondary Outcome: Part 1-Amount Excreted in Urine (Ae) of GSK3342830 in Urine
Description: Ae is defined as amount of drug GSK3342830, excreted in urine. Urine samples were collected pre-dose (within a 24-hr period before dosing, may begin on Day -1) and 0 to 4, 4 to 8, 8 to 12, 12 to 24, and 24 to 48 hrs post-dose. Log untransformed values for Ae have been presented.
Time Frame: as for outcome 14
Population: PK Parameter Population
Measure: Mean (Standard Deviation); unit: Milligram
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Milligram | 239.6 (38.250) | 558.7 (260.49) | 968.9 (216.28) | 1816 (189.65) | 3919 (117.58) | 5999 (413.23)

23. Secondary Outcome: Part 1:Dose Proportionality: AUC (0-t)
Description: Blood samples were collected at Day 1 (pre-dose, 0.5 hr, 1 hr, 1.25 hr, 1.5 hr, 2 hr, 3 hr, 3.5 hr, 4 hr, 4.5 hr, 5 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr, 24 hr, 36 hr, 48hr post-dose. Dose proportionality was assessed for AUC(0-inf) and Cmax after single dose administration. AUC(0-inf) was selected as the AUC exposure measure as it is the default AUC parameter for single dose administration and the observed data permitted its calculation.
Time Frame: as for outcome 14
Population: PK Parameter Population
Groups:
- GSK3342830 250 mg to 6000 mg: The data for healthy adult participants in all the cohorts starting from GSK3342830, cohort 250 to 6000 mg, were assessed. The participants had received escalated doses from 250 mg, 500 mg, 1000 mg, 2000 mg, 4000 mg, and 6000 mg. Each dose was administered as a single intravenous infusion for 1 hr on Day 1.
Arm/Group | GSK3342830 250 mg to 6000 mg
Number analyzed (Participants) | 0

24. Secondary Outcome: Part 1:Dose Proportionality: AUC (0-inf)
Description: Blood samples were collected at Day 1 (pre-dose, 0.5 hr, 1 hr, 1.25 hr, 1.5 hr, 2 hr, 3 hr, 3.5 hr, 4 hr, 4.5 hr, 5 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr, 24 hr, 36 hr, 48 hr post-dose. The data for estimate slope for log dose, has been reported.
Time Frame: as for outcome 14
Population: PK Parameter Population
Measure: Mean (Standard Error); unit: hour*microgram per milliliter
Arm/Group | GSK3342830 250 mg to 6000 mg
Number analyzed (Participants) | 36
hour*microgram per milliliter | 0.988 (0.0198)

25. Secondary Outcome: Part 1:Dose Proportionality: Cmax
Description: Blood samples were collected at Day 1 (pre-dose, 0.5 hr, 1 hr, 1.25 hr, 1.5 hr, 2 hr, 3 hr, 3.5 hr, 4 hr, 4.5 hr, 5 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr, 24 hr, 36 hr, 48hr post-dose. The data for estimate slope for log dose, has been reported.
Time Frame: as for outcome 14
Population: PK Parameter Population
Measure: Mean (Standard Error); unit: microgram per milliliter
Arm/Group | GSK3342830 250 mg to 6000 mg
Number analyzed (Participants) | 36
microgram per milliliter | 0.968 (0.0384)

26. Secondary Outcome: Part 2-AUC (0-inf) of GSK3342830
Description: AUC (0-inf), was defined as AUC extrapolated from time zero to infinity Day 1 at pre-dose (15 minutes) and 0.5 hr, 1 hr (end of infusion), 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hrs after start of infusion. Single pre-dose samples on mornings of Days 3, 6, 9, 12, and 13. Serial samples (Day 15) time points: pre-dose (15 minutes) and 0.5 hr, 1 (end of infusion), 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hrs after start of infusion. The untransformed values for AUC(0-inf) have been presented.
Time Frame: Pre-dose, and 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hr post-dose at Day 1. Pre-dose on Day 3, 6, 9, 12, and 13. Pre-dose, and 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hr post-dose at Day 15
Population: PK Parameter Population
Measure: Mean (Standard Deviation); unit: hour *microgram per milliliter
Arm/Group | GSK3342830 1000 mg TID
Number analyzed (Participants) | 11
hour *microgram per milliliter | 156.5 (24.756)

27. Secondary Outcome: Part 2-Cmax of GSK3342830
Description: Cmax was defined as the maximum concentration of drug GSK3342830, in plasma. It was collected at Day 1 at pre-dose (15 minutes) and 0.5 hr, 1 hr (end of infusion), 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hrs after start of infusion. Single pre-dose samples on mornings of Days 3, 6, 9, 12, and 13. Serial samples (Day 15) time points: pre-dose (15 minutes) and 0.5 hr, 1 (end of infusion), 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hrs after start of infusion.
Time Frame: Pre-dose, and 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hr, post-dose at Day 1. Pre-dose on Day 3, 6, 9, 12, and 13. Pre-dose, and 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hr post-dose at Day 15
Population: PK Parameter Population.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | GSK3342830 1000 mg TID
Number analyzed (Participants) | 11
microgram per milliliter | 60.25 (10.875)

28. Secondary Outcome: Part 2-Tmax of GSK3342830
Description: Tmax was defined as time required to achieve Cmax for drug GSK3342830, in plasma. It was collected at Day 1 at pre-dose (15 minutes) and 0.5 hr, 1 hr (end of infusion), 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hrs after start of infusion. Single pre-dose samples on mornings of Days 3, 6, 9, 12, and 13. Serial samples (Day 15) time points: pre-dose (15 minutes) and 0.5 hr, 1 (end of infusion), 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hrs after start of infusion.
Time Frame: Pre-dose, and 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 h post-dose at Day 1. Pre-dose on Day 3, 6, 9, 12, and 13. Pre-dose, and 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 h post-dose at Day 15
Population: PK Parameter Population
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | GSK3342830 1000 mg TID
Number analyzed (Participants) | 11
hour | 1.023 (0.0754)

29. Secondary Outcome: Part 2-Terminal t1/2 of GSK3342830 in Plasma
Description: t ½ is defined as the time required by the drug to reduce to half its quantity. Blood samples were collected at Day 1 at pre-dose (15 minutes) and 0.5 hr, 1 hr (end of infusion), 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hrs after start of infusion. Single pre-dose samples on mornings of Days 3, 6, 9, 12, and 13. Serial samples (Day 15) time points: pre-dose (15 minutes) and 0.5 hr, 1 (end of infusion), 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hrs after start of infusion.
Time Frame: as for outcome 28
Population: PK Parameter Population
Measure: Mean (Standard Deviation); unit: hour
Groups:
- GSK3342830 1000 mg TID: Healthy adult participants in this repeat dose escalation cohort were administered GSK3342830 dose, in Part 2 as 1000 mg, as a single IV infusion on Day 1, TID, IV infusions (approximately every 8 hours) on Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, and 14, and a single IV infusion on Day 15.
Arm/Group | GSK3342830 1000 mg TID
Number analyzed (Participants) | 11
hour | 2.171 (0.21459)

30. Secondary Outcome: Part 2-Total CL of GSK3342830 in Plasma
Description: The systemic CL is a PK measure of volume of plasma from which the drug is removed per unit time. The blood samples of 3 mL were collected at Day 1 at pre-dose (15 minutes) and 0.5 hr, 1 hr (end of infusion), 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hrs after start of infusion. Single pre-dose samples on mornings of Days 3, 6, 9, 12, and 13. Serial samples (Day 15) time points: pre-dose (15 minutes) and 0.5 hr, 1 (end of infusion), 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hrs after start of infusion.
Time Frame: as for outcome 26
Population: PK Parameter Population
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | GSK3342830 1000 mg TID
Number analyzed (Participants) | 11
Liter per hour | 6.552 (1.1567)

31. Secondary Outcome: Part 2- Vss of Distribution of GSK3342830 in Plasma
Description: Vss reflects the actual blood and tissue volume into which a drug is distributed and the relative binding of drug to protein in these spaces. The blood samples of 3 mL were collected at Day 1 at pre-dose (15 minutes) and 0.5 hr, 1 hr (end of infusion), 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hrs after start of infusion. Single pre-dose samples on mornings of Days 3, 6, 9, 12, and 13. Serial samples (Day 15) time points: pre-dose (15 minutes) and 0.5 hr, 1 (end of infusion), 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hrs after start of infusion.
Time Frame: as for outcome 28
Population: PK Parameter Population
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | GSK3342830 1000 mg TID
Number analyzed (Participants) | 11
Liter | 17.04 (3.2541)

32. Secondary Outcome: Part 2-Urinary Excretion Ratio Relative to Dose Feu (t1-t2) of GSK3342830
Description: The Feu has been reported from 0 to 4, 4 to 8, 8 to 12, 12 to 24 and 24 to 48 hrs. These were collected in opaque bottles at pre-dose (within a 24-hr period before dosing, may begin on Day -1) and 0 to 4, 4 to 8, 8 to 12, 12 to 24, and 24 to 48 hrs post-dose.
Time Frame: as for outcome 26
Population: PK Parameter Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles)
Measure: Mean (Standard Deviation); unit: Percentage of excretion ratio
Arm/Group | GSK3342830 1000 mg TID
Number analyzed (Participants) | 11
Percentage of excretion ratio
  Day 1 Feu (0-8), n=11 | 90.39 (5.9551)
  Day 1 Feu (8-24), n= 11 | 4.855 (1.3990)
  Day 15, Feu (0-8), n=6: number analyzed (Participants) | 6
  Day 15, Feu (0-8), n=6 | 89.80 (19.319)
  Day 15, Feu (8-24), n=6: number analyzed (Participants) | 6
  Day 15, Feu (8-24), n=6 | 4.530 (2.9358)

33. Secondary Outcome: Part 2- Trough Concentration (Ctau)
Description: Blood samples were collected on Pre-dose, and 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 h post-dose at Day 1. Pre-dose on Day 3, 6, 9, 12, and 13. Pre-dose, and 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 h post-dose at Day 15. The untransformed values for Ctau have been presented.
Time Frame: as for outcome 28
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | GSK3342830 1000 mg TID
Number analyzed (Participants) | 11
microgram per milliliter
  Day 1 (n=11) | 3.366 (0.82694)
  Day 15 (n=6): number analyzed (Participants) | 6
  Day 15 (n=6) | 3.059 (0.55052)

34. Secondary Outcome: Part 2-CLr of GSK3342830 in Urine
Description: The renal CLr is a PK measure of volume of plasma from which the drug is removed per unit time.These were collected in opaque bottles on Day 1 and Day 15 at (Pre-dose, 0 to 8 and 8 to 24 hrs post-dose). The untransformed values for CLr have been presented.
Time Frame: as for outcome 28
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | GSK3342830 1000 mg TID
Number analyzed (Participants) | 11
Liter per hour
  Day 1 (n=11) | 6.261 (1.3406)
  Day 15 (n=6): number analyzed (Participants) | 6
  Day 15 (n=6) | 6.174 (1.3504)

35. Secondary Outcome: Part 2- Ae of GSK3342830 in Urine
Description: Ae defines as the amount of drug GSK3342830, excreted in urine. These were collected in opaque bottles on Day 1 and Day 15 at (Pre-dose, 0 to 8 and 8 to 24 hrs post-dose). The untransformed values for Ae have been presented.
Time Frame: Day 1 and Day 15 at (Pre-dose, 0 to 8 and 8 to 24 hrs post-dose)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | GSK3342830 1000 mg TID
Number analyzed (Participants) | 11
milligram
  Day 1 (n=11) | 952.4 (61.274)
  Day 15 (n=6): number analyzed (Participants) | 6
  Day 15 (n=6) | 964.9 (223.30)

36. Secondary Outcome: Part 2: AUC From Time Zero to Last Measurable Concentration AUC (0- Tau)
Description: It was defined as Area Under the Concentration-time Curve From Time Zero (Pre-dose) to the time of the last measureable concentration. Blood samples were collected on Day 1 at indicated timepoints pre-dose, 0.5 hr, 1hr, 1.25 hr, 1.5 hr, 2 hr, 3 hr,3.5 hr, 4 hr, 4.5 hr, 5 hr, 6 hr, 8 hr, 10 hr, 12 hr, 16 hr 24 hr, 36 hr and 48 hr post-dose. Log untransformed values for AUC (0 to tau) have been presented.
Time Frame: as for outcome 14
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: hour*microgram per milliliter
Arm/Group | GSK3342830 1000 mg TID
Number analyzed (Participants) | 11
hour*microgram per milliliter
  Day 1 (n=11) | 145.6 (23.344)
  Day 15 (n=6): number analyzed (Participants) | 6
  Day 15 (n=6) | 156.1 (14.612)

37. Secondary Outcome: Part 2: Dose Proportionality: AUC (0-tau)
Description: Blood samples were collected at Pre-dose, and 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hr post-dose at Day 1. Pre-dose on Day 3, 6, 9, 12, and 13. Pre-dose, and 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 hr post-dose at Day 15. Data cannot be summarized because only 1 dose level studied so dose proportionality analysis cannot be performed as no comparison can be conducted.
Time Frame: as for outcome 27
Population: PK Parameter Population
Arm/Group | GSK3342830 1000 mg TID
Number analyzed (Participants) | 0

38. Secondary Outcome: Part 2: Observed Accumulation Ratio (Ro) Based on AUC and Cmax of GSK3342830 After Administration of Repeat IV Doses, as Data Permit
Description: The accumulation ratio has been reported. Sampling was done at Pre-dose, and 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 h post-dose at Day 1. Pre-dose on Day 3, 6, 9, 12, and 13. Pre-dose, and 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 h post-dose at Day 15. Data cannot be summarized because only 1 dose level studied so dose proportionality analysis cannot be performed as no comparison can be conducted.
Time Frame: as for outcome 28
Population: PK Parameter Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GSK3342830 1000 mg TID
Number analyzed (Participants) | 6
Ratio | 1.117 (0.16167)

39. Secondary Outcome: Part 2: Steady-state Ratio (Rss) of GSK3342830 to Assess Time Invariance, as Data Permit
Description: Sampling was done at Pre-dose, and 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 h post-dose at Day 1. Pre-dose on Day 3, 6, 9, 12, and 13. Pre-dose, and 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 h post-dose at Day 15. Since the study was terminated early, data is only available for one dose level for Part 2. Some subjects have only partial data and were not dosed on Day 15.
Time Frame: as for outcome 28
Population: PK Parameter Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GSK3342830 1000 mg TID
Number analyzed (Participants) | 6
Ratio | 1.033 (0.14336)

40. Secondary Outcome: Part 2: Trough Plasma Concentrations at the End of the Dosing Interval (Ctau) to Assess the Achievement of Steady-state of GSK3342830 After Administration of Repeat IV Doses, as Data Permit
Description: Sampling was done at Pre-dose, and 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 h post-dose at Day 1. Pre-dose on Day 3, 6, 9, 12, and 13. Pre-dose, and 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, and 8 h post-dose at Day 15. The untransformed values for Ctau have been presented.
Time Frame: as for outcome 28
Population: PK Parameter Population
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | GSK3342830 1000 mg TID
Number analyzed (Participants) | 11
microgram per milliliter
  Day 1 (n=11) | 3.366 (0.82694)
  Day 15 (n=6): number analyzed (Participants) | 6
  Day 15 (n=6) | 3.059 (0.55052)

ADVERSE EVENTS:
Time Frame: SAEs and AEs were collected from start of study treatment (Day 1) up to Day 56
Description: Safety population was used and on-treatment AEs and SAEs were reported.
Groups:
- GSK3342830 250 mg: Healthy adult participants in this cohort, were administered GSK3342830 dose in Part 1 as 250 mg,for 1 hr, as a single IV infusion, on Day 1.
Arm/Group | GSK3342830 250 mg | GSK3342830 500 mg | GSK3342830 1000 mg | GSK3342830 2000 mg | GSK3342830 4000 mg | GSK3342830 6000 mg | Placebo, Part 1 | GSK3342830 1000 mg TID | Placebo, Part 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/11 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/11 | 0/3
Other Adverse Events (participants affected / at risk) | 5/6 | 4/6 | 2/6 | 5/6 | 5/6 | 4/6 | 11/12 | 11/11 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK3342830 250 mg (N=6) | GSK3342830 500 mg (N=6) | GSK3342830 1000 mg (N=6) | GSK3342830 2000 mg (N=6) | GSK3342830 4000 mg (N=6) | GSK3342830 6000 mg (N=6) | Placebo, Part 1 (N=12) | GSK3342830 1000 mg TID (N=11) | Placebo, Part 2 (N=3)
Catheter site pain (General disorders) | 0 | 1 | 0 | 2 | 2 | 3 | 2 | 7 | 2
Application site dermatitis (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Application site reaction (General disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 1 | 1 | 2 | 1 | 6 | 7 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Catheter site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT02751424/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT02751424/SAP_001.pdf